CLINICAL TRIAL: NCT02417051
Title: The Efficacy of a Brief Resilience Training Program for Hurricane Sandy Disaster Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Northwell Health (Other); Rutgers University (Other); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Adam Gonzalez, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-HITEP-140021-01-00
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Psychological Stress
Keywords: Psychological Resilience; Perceived Stress; Psychological Stress; Disaster Worker; Superstorm Sandy; Mental Health; Prevention
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resiliency Training (Experimental): Intervention: Disaster Worker Resiliency Training (DWRT) Program.
  Interventions: Behavioral: Disaster Worker Resiliency Training
- Waitlist (No Intervention): Waitlist control: Participants to be offered the program after completion of the trial.

INTERVENTIONS:
Behavioral: Disaster Worker Resiliency Training — The Disaster Worker Resilience Training (DWRT) Program is a 4 hour program which consists of a participant training manual, an instructor-training manual, and a digital presentation. It uses adult training techniques that emphasize active participation in individual and group experiential learning activities. The curriculum is organized into a preface and four chapters, each with action oriented learning objectives. Overall program objectives include a demonstrate an ability to: 1) Recognize signs and symptoms of disaster work-related stress, 2) Obtain support through employer and community resources, and 3) Build resilience by using stress reduction and coping strategies.
  Other Names: Disaster Worker Resilience Training (DWRT) Program
  Arms: Resiliency Training

SUMMARY:
The goal of this project is to adapt and test the efficacy of the National Institute of Environmental Health and Safety (NIEHS) Disaster Worker Resilience Training (DWRT) Program for Superstorm Sandy responders. The DWRT is a brief, 4-5 hour training program designed to improve resilience for stress reactions in active emergency responders. A total of 120 participants will be recruited. 60 will receive the DWRT, and 60 will be assigned to a waitlist control condition. A three-month assessment period will be utilized to enable us to evaluate the effects of the intervention. Participants assigned to the waitlist condition will be offered the option to participant in the course following completion of the 3 month wait period. It is hypothesized that, participants attending the DWRT program, as compared to those in the waitlist condition, will show increased resilience at three months post-intervention as indicated by lower perceived stress, greater posttraumatic growth, more positive health behaviors (e.g., sleep, nutrition, exercise), and fewer new PTSD and depression symptoms. It is predicted that participants attending the DWRT program, as compared to those in the waitlist condition, will demonstrate greater awareness of the mental health effects of disasters, including the symptoms of PTSD and depression. It is predicted that, participants attending the DWRT program, as compared to those in the waitlist condition, will endorse more positive attitudes towards mental health care, including willingness to seek treatment if needed.

DETAILED DESCRIPTION:
This project is a scientific collaboration between the World Trade Center (WTC) Health Program at Stony Brook University (SBU), the Epidemiology Program at North Shore-LIJ Health System (NSLIJ), and Rutgers University. The goal is to adapt and test the efficacy of the National Institute of Environmental Health and Safety (NIEHS) Disaster Worker Resilience Training (DWRT) Program for Sandy responders by leveraging data from the ongoing projects and the expertise of collaborators at these sites. The DWRT program was originally designed for and piloted with responders to the 2010 Deep Water Horizon oil spill. Knowledge from the ongoing Sandy projects will be used to tailor this intervention to address Sandy-specific risk factors and unique features of the responder communities in the New York Metropolitan area. Responders identified from ongoing projects at SBU (N=1500, 50% anticipated eligible) and other current local disaster responders will be targeted for enrollment. The objectives are to: (1) to adapt the DWRT program for this population; (2) recruit and randomly assign responders (N = 120) to the DWRT program or a waitlist control condition; (3) assess the efficacy of this intervention to enhance resilience over a three month period; and (4) host forums with community stakeholders to share information on this program and its outcomes. The expected outcomes are: (1) efficacy data on the DWRT program, and (2) qualitative data on the acceptability of this intervention to Sandy responders. The products are: (1) a final report; (2) articles for publication; (3) abstracts for national conferences; and (4) a training manual, participant workbook, and presenter materials.

ELIGIBILITY:
Inclusion Criteria:

* Participated as a volunteer or professional in Hurricane Sandy relief efforts.
* Report that they are still an active disaster responder (i.e., they may be called upon to participate in future disaster relief efforts) as either a volunteer or professional.

Exclusion Criteria:

* An inability to comprehend the intervention in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | 3 months post-intervention
  Perceived Stress Scale (PSS; Cohen, Karmarck, and Mermelstein, 1983).

SECONDARY OUTCOMES:
Post-Traumatic Stress Disorder Symptoms | 3 months post-intervention
  PTSD Checklist for DSM-5 (PCL-5; Weathers, Litz, Keane, Palmieri, Marx, & Schnurr, 2013).
Depression Symptoms | 3 months post-intervention
  Patient Health Questionnaire-9 (PHQ-9; Spitzer, Kroenke, & Williams, 1999).
Mental Illness Stigma | 3 months post-intervention
  Attitudes Towards Mental Illness Questionnaire (ATMIQ).
Attitudes Towards Seeking Professional Help | 3 months post-intervention
  Attitudes Towards Seeking Professional Help Survey (ATSPH; Bacon, Fischer & Farina, 1995).
Post-traumatic Growth | 3 months post-intervention
  Post-Traumatic Growth Inventory-Short Form (PTGI-SF; Cann et al., 2010).
Health Promoting Behaviors | 3 months post-intervention
  Health Promoting Lifestyles Profile-II (HPLP-II; Walker, Sechrist, & Pender, 1995).

CONTACTS AND LOCATIONS:
Overall Officials: Adam Gonzalez, PhD, Principal Investigator — Stony Brook University

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Weathers, FW., Litz, BT, Keane, TM, Palmieri, PA, Marx, BP, & Schnurr, PP. The PTSD checklist for DSM-5 (PCL-5). National Center for PTSD. 2013.
- [Background] Cann A, Calhoun LG, Tedeschi RG, Taku K, Vishnevsky T, Triplett KN, Danhauer SC. A short form of the Posttraumatic Growth Inventory. Anxiety Stress Coping. 2010;23(2):127-37. doi: 10.1080/10615800903094273. PMID 19582640
- [Background] Fischer, Edward H, and Farina, A. Attitudes toward Seeking Professional Psychological Help: A Shortened Form and Considerations for Research. Journal of College Student Development 36(4): 368-73, 1995.
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860
- See also: Link to NIEHS Disaster Worker Training Program Materials — https://tools.niehs.nih.gov/wetp/index.cfm?id=2528